CLINICAL TRIAL: NCT01833572
Title: A Single-arm, Phase II Study of Preoperative Gefitinib for Stage II-IIIa NSCLC With Activating EGFR Mutation
Brief Title: Preoperative Gefitinib for EGFR Mutant II-IIIa NSCLC (ECTOP-1001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISSIRES0081; FUSCC1301 (Other: Fudan University Shanghai Cancer Center)
Record Dates: First submitted 2013-04-11; First posted 2013-04-17 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Non-small-cell Lung Cancer
Keywords: epidermal growth factor receptor; EGFR mutation; Tyrosine kinase inhibitor; gefitinib; neo-adjuvant therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

ARMS (1):
- Gefitinib (Experimental): A total of 42 cases of resectable stage II-IIIA NSCLCs patients with EGFR activating mutations will be enrolled in this arm.Gefitinib 250 mg/day oral daily is given to patients after enrolment for 42 days or until disease progression or unacceptable toxicity.
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — Eligible participants will be given orally gefitinib 250mg daily before surgery for 42 days or until disease progression or unacceptable toxicity. Best supportive care is allowed in this period.
  Other Names: Iressa

SUMMARY:
This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-1001. This is an open-label, single-arm, phase II interventional clinical trial. The investigators hypothesize that the application of EGFR-TKI, like gefitinib will be efficient and safe in a neo-adjuvant setting. 42 resectable stage II-IIIa NSCLC patients with EGFR activating (19/21) mutations will be eligible to be enrolled. EGFR mutation will be prospectively tested in all the participants' biopsy samples and confirmed in surgical resected samples. Eligible patients will be given gefitinib 250mg for 42days followed with surgical resection of tumor. Efficacy of preoperative gefitinib is based on radiographic (CT response/ORR), pathologic (pathologic response), surgical (complete resection) evaluations, and safety is based on adverse effect evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Pathologically confirmed non-small cell lung cancer with EGFR exon 19 deletion or exon 21 L858 mutation.
3. Clinically or pathologically confirmed stage II-IIIA
4. Tolerable to complete resection of lung cancer
5. Male or female aged 18 years and over
6. Able to comply with the required protocol and follow-up procedures, and able to receive oral medications
7. ECOG performance status 0-1.
8. Life expectancy ≥12 weeks.
9. Adequate hematological function: Absolute neutrophil count (ANC) ≥2.0 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
10. Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN); Aspartate amino transferase (AST) and alanine amino transferase (ALT) ≤ 2.5 x upper limit of normal (ULN).
11. Adequate renal function: Serum creatinine ≤ 1.5 x upper limit of normal (ULN), and creatinine clearance≥ 60 ml/min.
12. Measurable disease according to the preset criteria .

Exclusion Criteria:

1. Known severe hypersensitivity to gefitinib or any of the excipients of this product
2. Any serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study
3. Interstitial lung disease(ILD) or pulmonary fibrosis; impaired pulmonary function (e.g. FEV1 <40% predicted value, artery blood gas PaO2<60mmHg)
4. Patients with prior exposure to agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
5. Patients with prior exposure to chemotherapy, irradiation or systemic anti-cancer therapy (e.g. monoclonal antibody therapy) for lung cancer.
6. Previous or current malignancies of other histologies within the last 5 years with the exception of the following: other malignancies cured by surgery alone and having a continuous disease-free survival of 5 years; cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix.
7. Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within six months, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
8. Eye inflammation or eye infection not fully treated or predisposing factor of this.
9. Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the subject at high risk for treatment-related complications.
10. Patient who has serious active infection
11. Patients who harbouring exon 20 T790M mutation.
12. Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | at day 42 of gefitinib treatment

SECONDARY OUTCOMES:
Pathologic response rate | Pathologic response rate is depended on the pathology dignosis after surgery, an expected average of 8 weeks from enrollment.
Complete resection rate | Complete resection rate is depended on the pathology dignosis after surgery, an expected average of 8 weeks from enrollment.
Number of participants with adverse events | During the neoadjuvant and perioperative period, an expected average of 10 weeks from enrollment
Quality of life (QoL) | During the neoadjuvant period, an expected average of 6 weeks from enrollment
Disease free survival (DFS) | Participants after surgery will receive long-term follow-up for up to 5 years
Overall survival (OS) | Participants after surgery will receive long-term follow-up for up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, MD, Principal Investigator — Fudan Univerisity Shanghai Cancer Center
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Background] Goldstraw P, Crowley J, Chansky K, Giroux DJ, Groome PA, Rami-Porta R, Postmus PE, Rusch V, Sobin L; International Association for the Study of Lung Cancer International Staging Committee; Participating Institutions. The IASLC Lung Cancer Staging Project: proposals for the revision of the TNM stage groupings in the forthcoming (seventh) edition of the TNM Classification of malignant tumours. J Thorac Oncol. 2007 Aug;2(8):706-14. doi: 10.1097/JTO.0b013e31812f3c1a. PMID 17762336
- [Background] Rena O, Carsana L, Cristina S, Papalia E, Massera F, Errico L, Bozzola C, Casadio C. Lymph node isolated tumor cells and micrometastases in pathological stage I non-small cell lung cancer: prognostic significance. Eur J Cardiothorac Surg. 2007 Dec;32(6):863-7. doi: 10.1016/j.ejcts.2007.09.014. Epub 2007 Nov 1. PMID 17936004
- [Background] Gilligan D, Nicolson M, Smith I, Groen H, Dalesio O, Goldstraw P, Hatton M, Hopwood P, Manegold C, Schramel F, Smit H, van Meerbeeck J, Nankivell M, Parmar M, Pugh C, Stephens R. Preoperative chemotherapy in patients with resectable non-small cell lung cancer: results of the MRC LU22/NVALT 2/EORTC 08012 multicentre randomised trial and update of systematic review. Lancet. 2007 Jun 9;369(9577):1929-37. doi: 10.1016/S0140-6736(07)60714-4. PMID 17544497
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Zhou C, Wu YL, Chen G, Feng J, Liu XQ, Wang C, Zhang S, Wang J, Zhou S, Ren S, Lu S, Zhang L, Hu C, Hu C, Luo Y, Chen L, Ye M, Huang J, Zhi X, Zhang Y, Xiu Q, Ma J, Zhang L, You C. Erlotinib versus chemotherapy as first-line treatment for patients with advanced EGFR mutation-positive non-small-cell lung cancer (OPTIMAL, CTONG-0802): a multicentre, open-label, randomised, phase 3 study. Lancet Oncol. 2011 Aug;12(8):735-42. doi: 10.1016/S1470-2045(11)70184-X. Epub 2011 Jul 23. PMID 21783417
- [Background] Rizvi NA, Rusch V, Pao W, Chaft JE, Ladanyi M, Miller VA, Krug LM, Azzoli CG, Bains M, Downey R, Flores R, Park B, Singh B, Zakowski M, Heelan RT, Shen R, Kris MG. Molecular characteristics predict clinical outcomes: prospective trial correlating response to the EGFR tyrosine kinase inhibitor gefitinib with the presence of sensitizing mutations in the tyrosine binding domain of the EGFR gene. Clin Cancer Res. 2011 May 15;17(10):3500-6. doi: 10.1158/1078-0432.CCR-10-2102. Epub 2011 May 10. PMID 21558399
- [Background] Lara-Guerra H, Waddell TK, Salvarrey MA, Joshua AM, Chung CT, Paul N, Boerner S, Sakurada A, Ludkovski O, Ma C, Squire J, Liu G, Shepherd FA, Tsao MS, Leighl NB. Phase II study of preoperative gefitinib in clinical stage I non-small-cell lung cancer. J Clin Oncol. 2009 Dec 20;27(36):6229-36. doi: 10.1200/JCO.2009.22.3370. Epub 2009 Nov 2. PMID 19884551
- [Background] Schaake EE, Kappers I, Codrington HE, Valdes Olmos RA, Teertstra HJ, van Pel R, Burgers JA, van Tinteren H, Klomp HM. Tumor response and toxicity of neoadjuvant erlotinib in patients with early-stage non-small-cell lung cancer. J Clin Oncol. 2012 Aug 1;30(22):2731-8. doi: 10.1200/JCO.2011.39.4882. Epub 2012 Jul 2. PMID 22753915
- [Background] Haura EB, Sommers E, Song L, Chiappori A, Becker A. A pilot study of preoperative gefitinib for early-stage lung cancer to assess intratumor drug concentration and pathways mediating primary resistance. J Thorac Oncol. 2010 Nov;5(11):1806-14. doi: 10.1097/JTO.0b013e3181f38f70. PMID 20881637
- [Background] Lynch TJ, Bell DW, Sordella R, Gurubhagavatula S, Okimoto RA, Brannigan BW, Harris PL, Haserlat SM, Supko JG, Haluska FG, Louis DN, Christiani DC, Settleman J, Haber DA. Activating mutations in the epidermal growth factor receptor underlying responsiveness of non-small-cell lung cancer to gefitinib. N Engl J Med. 2004 May 20;350(21):2129-39. doi: 10.1056/NEJMoa040938. Epub 2004 Apr 29. PMID 15118073
- [Background] Scagliotti GV, Pastorino U, Vansteenkiste JF, Spaggiari L, Facciolo F, Orlowski TM, Maiorino L, Hetzel M, Leschinger M, Visseren-Grul C, Torri V. Randomized phase III study of surgery alone or surgery plus preoperative cisplatin and gemcitabine in stages IB to IIIA non-small-cell lung cancer. J Clin Oncol. 2012 Jan 10;30(2):172-8. doi: 10.1200/JCO.2010.33.7089. Epub 2011 Nov 28. PMID 22124104